CLINICAL TRIAL: NCT02981264
Title: Transcricoid Injection vs. Spray as You go Method for Local Anaesthesia During Endobronchial Ultrasound-guided Transbronchial Needle Aspiration (EBUS-TBNA): A Randomised Controlled Trial
Brief Title: Transcricoid Injection vs. Spray as You go Method for Local Anaesthesia During EBUS-TBNA
Acronym: CRISPEN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: All India Institute of Medical Sciences (Other)
Responsible Party: Principal Investigator, Karan Madan, Dr. Karan Madan, MD, DM Assistant Professor, Pulmonary Medicine and Sleep Disorders, All India Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: Transcricoid EBUS RCT
Record Dates: First submitted 2016-12-01; First posted 2016-12-05 (Estimated); Last update posted 2020-11-30 (Actual); Status verified 2020-11

CONDITIONS: Pulmonary Disease
Keywords: Bronchoscopy; Lignocaine; Endobronchial Ultrasound
MeSH Terms: conditions — Lung Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Transcricoid (Active Comparator): Lignocaine delivery using transcricoid injection
  Interventions: Drug: Transcricoid Injection
- Spray as You go (Active Comparator): Lignocaine delivery using spray as you go method
  Interventions: Drug: Spray as you go

INTERVENTIONS:
Drug: Transcricoid Injection
  Other Names: Lignocaine delivered through the cricothyroid membrane
  Arms: Transcricoid
Drug: Spray as you go
  Other Names: Lignocaine delivered through the bronchoscope working channel.
  Arms: Spray as You go

SUMMARY:
Endobronchial Ultrasound Guided Transbronchial Needle Aspiration (EBUS -TBNA) is commonly performed for diagnosis of mediastinal pathologies. The procedure can either be performed under general anaesthesia or under moderate sedation with topical anaesthesia. Most patients tolerate the procedure well although cough is often reported as a distressing symptom. Topical lignocaine is administered during endobronchial ultrasound for local anaesthesia. There is limited literature on the efficacy of transtracheal/transcricoid injection versus spray as you go method for lignocaine delivery to the airways during EBUS-TBNA. This study would help to determine the procedure comfort for the patient while using the transtracheal/transcricoid method vs the spray as you go method.

DETAILED DESCRIPTION:
For all patients meeting the inclusion criteria, the demographic profile including age, sex, weight, smoking history shall be recorded. A written informed consent will be obtained from all participants. The patients who undergo EBUS-TBNA under moderate sedation would be randomised in a one is to one ratio either to transcricoid injection or spray as you go lignocaine group. Prior to EBUS-TBNA, Blood pressure, pulse rate, respiratory rate and pulse oximetry saturation will be recorded at the baseline Patients in both the groups shall be prepared in a similar fashion except for the use of transcricoid injection in one group.

During the procedure, 2 ml aliquots of 1% lignocaine solution will be delivered through the bronchoscope when using spray-as-you go technique. Patients in the transcricoid group shall initially receive 5 ml of 2% lignocaine solution and additional aliquots of 1% lignocaine using the spray as you go method. The total lignocaine dose during the procedure will be recorded. The patients would be monitored for any adverse effects throughout the procedure. The bronchoscopist doing the procedure will be provided VAS charts to mark the severity of cough and overall procedure satisfaction. An audio recorder shall be used to record the cough count during the entire procedure.

Post procedure, patients will record the pain experienced while undergoing the procedure on the VAS scale.

ELIGIBILITY:
Inclusion Criteria:

* Indication for EBUS TBNA
* Age > 18 years

Exclusion Criteria:

* Refusal of consent
* Known documented hypersensitivity to lignocaine
* Procedure performed under general anaesthesia
* Pregnancy
* Hypoxemia (oxygen saturation [by pulse oximetry] < 92% with Fio2 of ≥ 0.3
* Bronchoscopy done through endotracheal or tracheostomy tube
* Midline neck mass or thyroid enlargement making the identification of
* cricothyroid membrane difficult'
* Patients with central airway obstruction
* Patients with active ongoing hemoptysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 365 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Overall cough count | At study completion approximately 12 months
  Cough count till reaching carina
Operator rated overall procedure satisfaction | Through study completion, an average of 1 year
  Operator rated satisfaction on VAS scale

SECONDARY OUTCOMES:
Time from scope insertion to crossing the vocal cords | At study completion approximately 12 months
  Time in seconds
Overall procedure duration | At study completion approximately 12 months
  Time in minutes
Total Lignocaine dose | At study completion approximately 12 months
  Total dose of lignocaine in milligrams

CONTACTS AND LOCATIONS:
Overall Officials: Randeep Guleria, MD, DM, Study Chair — All India Institute of Medical Sciences
Locations (1):
- AIIMS, New Delhi, India

IPD SHARING:
Plan to Share IPD: Yes
The data on demographics and outcomes shall be available on reasonable request
Time Frame: For two years since the study completion
Access Criteria: Available on reasonable request

REFERENCES:
- [Derived] Mittal S, Gupta N, Iyer H, Biswal SK, Tiwari P, Hadda V, Mohan A, Guleria R, Madan K. The cricothyroid versus Spray-As-You-Go method for topical anesthesia during Endobronchial Ultrasound-guided Transbronchial Needle Aspiration (EBUS-TBNA): The CRISPEN randomized clinical trial. Lung India. 2021 May-Jun;38(3):223-228. doi: 10.4103/lungindia.lungindia_801_20. PMID 33942745